CLINICAL TRIAL: NCT07280624
Title: Clinical Significance of Real Time PCR Panel in Children With Acute Gastrointestinal Symptoms
Brief Title: Diagnostic PCR Panel in Children With Acute Gastrointestinal Symptoms
Acronym: RealCAGI RCT
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Oulu (Other)
Collaborators: Oulu University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: OULU_EETTMK_39_2025
Record Dates: First submitted 2025-11-17; First posted 2025-12-12 (Actual); Last update posted 2025-12-12 (Actual); Status verified 2025-11

CONDITIONS: Gastroenteritis Acute; Gastrointestinal Symptoms; Abdominal Pain/ Discomfort; Vomiting in Infants and/or Children
Keywords: Multiplex PCR; Fecal samples; Diagnostic stewardship; Diarrhea; Vomiting; Abdominal pain; Gastrointestinal symptoms; Pediatrics; Children; Emergency department
MeSH Terms: conditions — Diarrhea; Vomiting; Abdominal Pain; Emergencies

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention: Rapid diagnostics group (Other): Immediate use of multiplex PCR panel for fecal samples
  Interventions: Diagnostic Test: Multiplex PCR gastrointestinal panel
- Control group (No Intervention): Control group without immediate multiplex PCR for fecal samples

INTERVENTIONS:
Diagnostic Test: Multiplex PCR gastrointestinal panel — Intervention includes a rapid use of multiplex PCR panel for gastrointestinal pathogens of fecal samples from children with acute gastrointestinal symptoms evaluated at a pediatric emergency room
  Other Names: Multiplex PCR of fecal samples
  Arms: Intervention: Rapid diagnostics group

SUMMARY:
This investigator-initiated randomized controlled trial compares the clinical impact of real time PCR of fecal samples in children with acute gastrointestinal symptoms at a pediatric emergency room. Specifically, the trial compares immediate testing of fecal samples using a multiplex PCR panel to a a control group with delayed test results.

DETAILED DESCRIPTION:
Acute gastroenteritis is one of the most common reasons for pediatric emergency visits in both general and pediatric emergency departments. For most of the children rehydration is the only therapy needed. However, a range of bacterial pathogens and parasites may need accurate diagnosis and targeted antimicrobial therapy. Use of molecular multiplex testing has increased detection of pathogens in children with acute gastrointestinal symptoms. The PCR tests currently available enable rapid identification of gastrointestinal pathogens, with the test results often being available during the day sample was taken. However, it is unclear which of the patients are most likely to benefit from testing. Also, there is considerable uncertainty about the cost-effectiveness of the multiplex panels used to test for suspected infectious gastroenteritis in hospital and community settings. The previous study by the research group demonstrated that acute gastrointestinal symptoms are one of the most common diagnoses and a major cost in high-income population.

The main hypothesis of the study is that real time multiplex PCR testing for gastrointestinal pathogens at pediatric emergency department setting could provide clinical benefit by allowing 1) earlier initiation of appropriate antimicrobial treatment, 2) reduce use of unnecessary antimicrobial treatment and 3) improve identification of conditions in need for follow-up.

To estimate the usefulness of real time multiplex PCR testing, an investigator-driven academic randomized (1:1) controlled trial will be conducted at the Pediatric Emergency Department of Oulu University Hospital, Finland. For eligibility, children aged under 16 years arriving to pediatric emergency due to acute gastrointestinal symptoms will be assessed. After obtaining the written consent, fecal specimens will be collected by the nurses from the first stool after arriving to hospital.

Multiplex PCR detects 13 gastrointestinal bacterial pathogens, 5 viral pathogens ands 4 parasitic species. QIAStat-Dx gastrointestinal panel 2 will be used.

The trial will compare two groups:

1. Intervention group will be tested by a relay-time PCR panel as soon as the fecal sample will arrive in the laboratory and the results will be given to the clinical physicians
2. Control group will undergo similar sampling as the intervention group but the results will be made available after 72 hours of sampling.

The composite primary outcome consists of three outcomes which are evaluated using medical records: 1) correctly targeted antimicrobial treatment, 2) untargeted antimicrobial treatment and 3) identification of conditions that require specific follow-up such as shiga-toxin producing EHEC.

Secondary outcomes, evaluated by medical records and electronic survey sent to families two weeks after the study visit, include: proportion of correctly targeted antimicrobial treatment, proportion of untargeted antimicrobial treatment, proportion of conditions in need for hospitalization or specific follow-up, time needed for clinician to receive the results of the samples, length of hospital stay, time to correct diagnosis, resolution of symptoms, laboratory and radiology costs, total costs, need for surgical consultation and proportion of patients needing surgical procedure, proportion of unscheduled revisits and proportion of correctly used hospital infection control measures.

ELIGIBILITY:
Inclusion Criteria:

* Child or adolescent < 16 years of age
* Visiting pediatric ED
* Presence of gastrointestinal symptom or symptoms (diarrhea, vomiting or abdominal pain)

Exclusion Criteria:

* Need of cardiopulmonary resuscitation at the ED
* Need of immediate transfer to the intensive care unit
* Hemato-oncological disease
* Severe immunosuppression
* Bloody diarrhea
* Clinical suspicion of typhoid/paratyphoid fever

Max Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 526 (Estimated)
Dates: Start 2025-12-15 (Estimated); Primary Completion 2027-12-15 (Estimated); Study Completion 2028-02-15 (Estimated)

PRIMARY OUTCOMES:
Impact on clinical decision making | 72 hours from initial contact at the ED
  Primary outcome comprises the proportion of participants with 1) targeted antimicrobial therapy based on PCR results 2) untargeted antimicrobial therapy avoided based on PCR result, OR 3) specific clinical follow up planned based on PCR result, namely EHEC infection

SECONDARY OUTCOMES:
Proportion of children with correctly targeted antimicrobial therapy | 72 hours from initial contact at the ED
  Proportion of children with correctly targeted antimicrobial therapy based on PCR results
Proportion of children needing hospitalization or specific follow up | 72 hours from initial contact at the ED
  Proportion of children needing hospitalization or specific follow up
Time to receive the laboratory results | 7 days from the initial presentation to the ED
  Time (hours) from the initial presentation at the ED to the laboratory results given to the clinicians
Length of stay | 30 days from the presentation to the ED
  Length of hospital stay, time (hours) before discharge
Time to correct diagnosis | 30 days from the initial presentation at the ED
  Time (hours) for the most probable correct diagnosis after the presentation at the ED
Time to resolution of symptoms | 28 days
  The time (days) to the resolution of gastrointestinal symptoms based on medical record review and parental electronic survey at 2 weeks and 4 weeks after initial visit
The overall cost of diagnostic procedures | 72 hours from the initial contact
  The cost (euros) per participant including all laboratory and radiological costs, adding the cost of multiplex PCR for the intervention group
Total cost of treatment | 30 days from the initial presentation
  The total cost of treatment including hospital stay, and visits at ED
Need for a surgical consultation | 72 hours from initial presentation
  The proportion of children needing a surgical consultation
Surgical operation | 72 hours from the initial presentation
  The proportion of children undergoing abdominal surgery or operation
Revisit at the ED | 30 days
  Proportion of participants with revisits to the ED
Correct hospital isolation measures | 72 hours from initial presentation
  The proportion of children placed in a correct way in an infectious diseases ward due to a nosocomially problematic pathogen such as norovirus
Correct use of personal protective equipment | 72 hours from the initial presentation
  The proportion of participants treated correctly using personal protective equipment based on multiplex PCR findings
Pediatric infectious diseases consultation | 72 hours after the initial presentation at the ED
  The proportion of participants needing a pediatric infectious diseases consultation

CONTACTS AND LOCATIONS:
Overall Officials: Terhi S Ruuska-Loewald, MD, PhD, Principal Investigator — Oulu University Hospital and University of Oulu

IPD SHARING:
Plan to Share IPD: Yes
The individual participant data on the primary outcome of participants according to groups. No identifying participant data will be shared according to EU GDPR regulations. Study protocol and statistical analysis plan will be hared upon submission of the manuscript.
Supporting Information: Study Protocol, SAP
Time Frame: Upon the submission of the manuscript

REFERENCES:
- [Background] Poyry H, Kiviniemi M, Raappana A, Honkila M, Paalanne N, Pokka T, Valmari P, Renko M, Tapiainen T. The most common diagnoses and costs of paediatric emergency department visits: A population-based cohort study. Acta Paediatr. 2022 Jan;111(1):169-170. doi: 10.1111/apa.16087. Epub 2021 Sep 20. No abstract available. PMID 34448253
- [Background] Freeman K, Mistry H, Tsertsvadze A, Royle P, McCarthy N, Taylor-Phillips S, Manuel R, Mason J. Multiplex tests to identify gastrointestinal bacteria, viruses and parasites in people with suspected infectious gastroenteritis: a systematic review and economic analysis. Health Technol Assess. 2017 Apr;21(23):1-188. doi: 10.3310/hta21230. PMID 28619124

DOCUMENTS (1):
  • Study Protocol (2025-10-16): https://cdn.clinicaltrials.gov/large-docs/24/NCT07280624/Prot_000.pdf